CLINICAL TRIAL: NCT00047138
Title: Nephroblastoma (Wilms Tumour) Clinical Trial And Study
Brief Title: Chemotherapy Before and After Surgery in Treating Children With Wilm's Tumor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: Societe Francaise Oncologie Pediatrique (Other); Children's Cancer and Leukaemia Group (Other); German Society for Pediatric Oncology and Hematology GPOH gGmbH (Other)
Responsible Party: Sponsor
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000257531; SIOP-WT-2001; SFOP-SIOP-WT-2001; CCLG-SIOP-WT-2001; GPOH-GERMANY-SIOP-WT-2001; EU-20208
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Kidney Cancer
Keywords: blastema predominant Wilms tumor; epithelial predominant Wilms tumor; mixed cell type Wilms tumor; stage I Wilms tumor; stage II Wilms tumor; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor; stromal predominant Wilms tumor
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Dactinomycin; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Vincristine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Biological: dactinomycin
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: vincristine sulfate
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving combination chemotherapy before surgery may shrink the tumor so it can be removed during surgery. Giving more chemotherapy after surgery may kill any remaining tumor cells. It is not yet known which chemotherapy regimen after surgery is most effective in treating Wilm's tumor.

PURPOSE: Phase III trial to study the effectiveness of chemotherapy before and after surgery in treating children who have Wilm's tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in children with Wilms' tumor treated with pre-operative chemotherapy.
* Compare the response rate in children with intermediate-risk stage II or III Wilms' tumor treated with or without doxorubicin after surgery.
* Determine the prognostic significance of histological subtypes in these patients after pre-operative chemotherapy.
* Determine whether reduced treatment minimizes acute and late toxicity without jeopardizing event-free and overall survival in patients with focal anaplasia or intermediate-risk stage I Wilms' tumor.
* Determine the prognostic significance of tumor volume and specimen weight after pre-operative chemotherapy and its relation to histological subtype in these patients.
* Determine the effect of single-dose dactinomycin as pre-operative chemotherapy in these patients.
* Correlate allele loss at 16q, 1p, and other chromosomal regions with relapse-free and overall survival of patients treated with these regimens.
* Correlate allele losses with clinical risk factors (e.g., histological appearance and tumor volume) after pre-operative chemotherapy in these patients.
* Determine laboratory indicators of myocardial damage in patients treated with these regimens.
* Determine the prognostic significance of the percentage of necrosis after pre-operative chemotherapy, in terms of type and amount of residual viable tumor, in these patients.

OUTLINE: This is a partially randomized, multicenter study. Patients are stratified according to country and participating center. Patients with intermediate-risk stage II or III disease are further stratified according to histology (blastemal vs epithelial vs stromal vs mixed).

Patients with localized disease receive neoadjuvant therapy comprising vincristine IV on days 1, 8, 15, and 22 and dactinomycin IV on days 1 and 15.

Patients undergo surgery during weeks 5 or 6.

Patients with low-risk stage I disease receive no further therapy.

Adjuvant chemotherapy begins after surgery and within 21 days of last dose of neoadjuvant chemotherapy.

Patients with intermediate-risk stage I disease receive vincristine IV on days 1, 8, 15, and 22 and dactinomycin IV on day 7.

Patients with intermediate-risk stage II or III disease are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive vincristine IV weekly for 8 weeks and then on days 1 and 7 of weeks 11, 14, 17, 20, 23, and 26. Patients also receive dactinomycin IV weekly on weeks 2, 5, 8, 11, 14, 17, 20, 23, and 26 and doxorubicin IV over 4-6 hours weekly on weeks 2, 8, 14, 20, and 26.
* Arm II: Patients receive vincristine and dactinomycin as in arm I. Patients with high-risk stage I disease receive chemotherapy as in arm I. Patients with low-risk stage II disease receive chemotherapy as in arm II.

Patients with high-risk stage II or III disease receive cyclophosphamide IV over 1 hour on days 1-3 and doxorubicin IV over 4-6 hours on day 1 on weeks 1, 7, 13, 19, 25, and 31. Patients also receive etoposide IV over 4 hours and carboplatin IV over 1 hour on days 1-3 on weeks 4, 10, 16, 22, 28, and 34.

Patients with intermediate-risk stage III or high-risk stage II or III disease also undergo radiotherapy for approximately 3 weeks during chemotherapy.

Patients with metastatic disease receive neoadjuvant chemotherapy comprising vincristine IV on day 1 of weeks 1-6, dactinomycin IV on day 1 of weeks 1, 3, and 5, and doxorubicin IV over 4-6 hours on day 1 of weeks 1 and 5.

Patients undergo surgery during week 7.

Within 2 weeks of surgery patients receive 1 of the following adjuvant chemotherapy regimens:

* Regimen A (no metastases or completely resected): Patients receive vincristine IV weekly for 8 weeks and then on weeks 11, 12, 14, 15, 17, 18, 20, 21, 23, 24, 26, and 27. Patients also receive dactinomycin IV on day 1 of weeks 2, 5, 8, 11, 14, 17, 20, 23, and 26 and doxorubicin IV over 4-6 hours on weeks 2, 8, 14, and 20. Some patients also undergo radiotherapy concurrently with chemotherapy for approximately 3 weeks.
* Regimen B (multiple inoperable metastases, incomplete resection, or high-risk primary disease): Patients receive etoposide IV over 4 hours and carboplatin IV over 1 hour on days 1-3 of weeks 4, 10, 13, 16, 22, 25, 28, and 34. Patients also receive cyclophosphamide IV over 1 hour on days 1-3 and doxorubicin IV over 4-6 hours on day 1 of weeks 1, 7, 19, and 31. Some patients also undergo radiotherapy concurrently with chemotherapy for approximately 3 weeks.

Patients are followed every 2-3 months for 2 years, every 3-6 months for 1-2 years, and then every 6-12 months thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 350 patients (174 per treatment arm) will be accrued for the randomized portion of this study within 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following:

  * Localized disease

    * Unilateral tumor
    * Histologically confirmed Wilms' tumor OR
    * Clinical and ultrasonic characteristics of nephroblastoma
    * No metastasis
    * Age 6 months to 17 years at diagnosis
    * No prior anticancer therapy
  * Metastatic disease

    * Unilateral tumor
    * Histologically confirmed Wilms' tumor OR
    * Clinical and ultrasonic characteristics of nephroblastoma
    * Age 18 and under
    * No prior anticancer therapy
  * Simultaneous bilateral tumors

    * No metastases
* No recurrent disease
* No other renal tumors

PATIENT CHARACTERISTICS:

Age

* See Disease Characteristics
* 18 and under

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No social or geographical reasons that would preclude study
* No other associated pathology that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy

Surgery

* No prior surgery
* No requirement for emergency or immediate surgery for any reason

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2001-01

PRIMARY OUTCOMES:
Event-free survival
Treatment failure, in terms of disease recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: Jan DeKraker, MD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Francois Pein, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris; Kathy Pritchard-Jones, MD, Study Chair — Royal Marsden NHS Foundation Trust; Norbert Graf, Study Chair — Universitaetsklinikum des Saarlandes
Locations (4):
- Institut Gustave Roussy, Villejuif, France
- Universitaetsklinikum des Saarlandes, Homburg, Germany
- Academisch Medisch Centrum at University of Amsterdam, Amsterdam, Netherlands
- Royal Marsden - Surrey, Sutton, England, United Kingdom

REFERENCES:
- [Background] Warmann SW, Nourkami N, Fruhwald M, Leuschner I, Schenk JP, Fuchs J, Graf N. Primary lung metastases in pediatric malignant non-Wilms renal tumors: data from SIOP 93-01/GPOH and SIOP 2001/GPOH. Klin Padiatr. 2012 Apr;224(3):148-52. doi: 10.1055/s-0032-1304600. Epub 2012 Apr 18. PMID 22513793
- [Background] Furtwangler R, Nourkami N, Alkassar M, von Schweinitz D, Schenk JP, Rube C, Siemer S, Leuschner I, Graf N. Update on relapses in unilateral nephroblastoma registered in 3 consecutive SIOP/GPOH studies - a report from the GPOH-nephroblastoma study group. Klin Padiatr. 2011 May;223(3):113-9. doi: 10.1055/s-0031-1275293. Epub 2011 Apr 20. PMID 21509706
- [Background] van den Heuvel-Eibrink MM, van Tinteren H, Rehorst H, Coulombe A, Patte C, de Camargo B, de Kraker J, Leuschner I, Lugtenberg R, Pritchard-Jones K, Sandstedt B, Spreafico F, Graf N, Vujanic GM. Malignant rhabdoid tumours of the kidney (MRTKs), registered on recent SIOP protocols from 1993 to 2005: a report of the SIOP renal tumour study group. Pediatr Blood Cancer. 2011 May;56(5):733-7. doi: 10.1002/pbc.22922. Epub 2010 Dec 22. PMID 21370404
- [Background] Warmann SW, Furtwangler R, Blumenstock G, Armeanu S, Nourkami N, Leuschner I, Schenk JP, Graf N, Fuchs J. Tumor biology influences the prognosis of nephroblastoma patients with primary pulmonary metastases: results from SIOP 93-01/GPOH and SIOP 2001/GPOH. Ann Surg. 2011 Jul;254(1):155-62. doi: 10.1097/SLA.0b013e318222015e. PMID 21670612
- [Background] Szavay P, Luithle T, Graf N, Furtwangler R, Fuchs J. Primary hepatic metastases in nephroblastoma--a report of the SIOP/GPOH Study. J Pediatr Surg. 2006 Jan;41(1):168-72; discussion 168-72. doi: 10.1016/j.jpedsurg.2005.10.021. PMID 16410128
- [Result] Smets AM, van Tinteren H, Bergeron C, De Camargo B, Graf N, Pritchard-Jones K, de Kraker J. The contribution of chest CT-scan at diagnosis in children with unilateral Wilms' tumour. Results of the SIOP 2001 study. Eur J Cancer. 2012 May;48(7):1060-5. doi: 10.1016/j.ejca.2011.05.025. Epub 2011 Jun 22. PMID 21703848
- [Result] Williams RD, Al-Saadi R, Chagtai T, Popov S, Messahel B, Sebire N, Gessler M, Wegert J, Graf N, Leuschner I, Hubank M, Jones C, Vujanic G, Pritchard-Jones K; Children's Cancer and Leukaemia Group; SIOP Wilms' Tumour Biology Group. Subtype-specific FBXW7 mutation and MYCN copy number gain in Wilms' tumor. Clin Cancer Res. 2010 Apr 1;16(7):2036-45. doi: 10.1158/1078-0432.CCR-09-2890. Epub 2010 Mar 23. PMID 20332316
- [Result] Messahel B, Williams R, Ridolfi A, A'hern R, Warren W, Tinworth L, Hobson R, Al-Saadi R, Whyman G, Brundler MA, Kelsey A, Sebire N, Jones C, Vujanic G, Pritchard-Jones K; Children's Cancer and Leukaemia Group (CCLG). Allele loss at 16q defines poorer prognosis Wilms tumour irrespective of treatment approach in the UKW1-3 clinical trials: a Children's Cancer and Leukaemia Group (CCLG) Study. Eur J Cancer. 2009 Mar;45(5):819-26. doi: 10.1016/j.ejca.2009.01.005. Epub 2009 Feb 21. PMID 19231157
- [Derived] Sudour-Bonnange H, van Tinteren H, Ramirez-Villar GL, Godzinski J, Irtan S, Gessler M, Chowdhury T, Audry G, Fuchs J, Powis M, van de Ven CP, Okoye B, Smeulders N, Vujanic GM, Verschuur A, L'Hermine-Coulomb A, de Camargo B, de Aguirre Neto JC, Schenk JP, van den Heuvel-Eibrink MM, Pritchard-Jones K, Graf N, Bergeron C, Furtwangler R. Characteristics and outcome of synchronous bilateral Wilms tumour in the SIOP WT 2001 Study: Report from the SIOP Renal Tumour Study Group (SIOP-RTSG). Br J Cancer. 2024 Oct;131(6):972-981. doi: 10.1038/s41416-024-02799-0. Epub 2024 Jul 30. PMID 39080350